CLINICAL TRIAL: NCT00865514
Title: Pharmacotoxicology of Trichloroethylene Metabolites: Short-term Effect of DCA on in Vivo Tyrosine Catabolism and MAAI Expression
Brief Title: Pharmacotoxicology of Trichloroethylene Metabolites
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in obtaining the solution from the compounding pharmacies caused a two year delay in start-up; the funding ended prior to study completion.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14617-CP-001; 5R01ES014617 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: dichloroacetate; tyrosine; maleylacetoacetate; trichloroethylene; leucine; haplotype
MeSH Terms: interventions — Dichloroacetic Acid; Leucine; Tyrosine; Genotype; Genes; Haplotypes; Amino Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Haplotypes and DCA metabolism (Experimental): Healthy men and women with different haplotypes will receive an infusion of leucine and tyrosine. The following day they begin a 5 day course of dichloroacetate (DCA)at a dose of 2.5mcg/kg/day. On day 6 they return and receive another infusion of leucine and tyrosine. After a 30 day washout period the subject returns and again receives an infusion of leucine and tyrosine. Then on day 2 they begin a dose of DCA at 25mg/kg for 5 days and then return for the final infusion of leucine and tyrosine.
  Interventions: Drug: Dichloroacetate; Genetic: Genotyping; Other: Leucine; Other: tyrosine

INTERVENTIONS:
Drug: Dichloroacetate — Healthy men and women with different haplotypes will receive an infusion of leucine and tyrosine. The following day they begin a 5 day course of dichloroacetate (DCA)at a dose of 2.5mcg/kg/day. On day 6 they return and receive another infusion of leucine and tyrosine. After a 30 day washout period the subject returns and again receives an infusion of leucine and tyrosine. Then on day 2 they begin a dose of DCA at 25mg/kg for 5 days and then return for the final infusion of leucine and tyrosine.
  Other Names: DCA; Leucine; Tyrosine
Genetic: Genotyping — Subjects will have 5 mls of blood drawn for genotyping
  Other Names: gene; haplotype
Other: Leucine — Healthy men and women with different haplotypes will receive an infusion of leucine and tyrosine. The following day they begin a 5 day course of dichloroacetate (DCA)at a dose of 2.5mcg/kg/day. On day 6 they return and receive another infusion of leucine and tyrosine. After a 30 day washout period the subject returns and again receives an infusion of leucine and tyrosine. Then on day 2 they begin a dose of DCA at 25mg/kg for 5 days and then return for the final infusion of leucine and tyrosine.
  Other Names: amino acid
Other: tyrosine — Healthy men and women with different haplotypes will receive an infusion of leucine and tyrosine. The following day they begin a 5 day course of dichloroacetate (DCA)at a dose of 2.5mcg/kg/day. On day 6 they return and receive another infusion of leucine and tyrosine. After a 30 day washout period the subject returns and again receives an infusion of leucine and tyrosine. Then on day 2 they begin a dose of DCA at 25mg/kg for 5 days and then return for the final infusion of leucine and tyrosine.
  Other Names: amino acid

SUMMARY:
This project focuses on the kinetics, metabolism and human toxicology of dichloroacetate (DCA)and tyrosine catabolism. The hypothesis is that tyrosine metabolism will be greatest in subject who harbor the KRT variant for GSTz1/MAAI for which DCA exhibits a high Km.

DETAILED DESCRIPTION:
Specific Aim 4. Quantify the effects of DCA on human tyrosine metabolism and on its own biotransformation in relation to dose and genotype.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective surgery for benign liver disease.
* Normal EKG and history
* Normal baseline labs

Exclusion Criteria:

* Pregnancy
* severe anemia, defined as a hematocrit < 30%.
* diabetes mellitus
* renal insufficiency, defined as a serum creatinine > 1.5 mg/dl or a creatinine clearance < 60 ml/min
* elevated liver enzymes
* psychiatric illness requiring medication
* primary biliary cirrhosis or any other form of cirrhosis
* viral hepatitis or non-viral steatohepatitis
* coronary heart disease, defined as requiring daily administration of anti-anginal drugs or as New York Heart Association Class III or IV heart failure
* malignancy of any type in any anatomical location

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Stacpoole, PhD, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] National Toxicology Program. Toxicology Carcinogenesis Studies of Trichloroethylene (Without Epichlorohydon)(CAS No. 7.9-011-6) in F3dd/N Rats B6C3F1 Mice (Gavage Studies). Research Triangle Park, NC: US Department of Health Human Services; Technical report series No. 243; NIH Publication 9:0-1779, 1990.
- [Background] LARC Monogr Eval Carcinog Risks Hum 11:263-276,1979.
- [Background] Page NN. Assessment of trichloroethylene as an occupational carcinogen. IARC Sci Publ (1971). 1979;(25):75-9. PMID 457166
- [Background] Federal Register 40(203):49032-49045, 1975.
- [Background] Westrick JJ, Mello JW, Thomas RF. The groundwater supply survey. J Am Water Works 76:52, 1984.
- [Background] Josephson J. ES Views: Implementing Superfund. Environ Sci Technol. 1986 Jan 1;20(1):23-8. doi: 10.1021/es00143a601. No abstract available. PMID 22300147
- [Background] Brown LP, Farrar DG, de Rooij CG. Health risk assessment of environmental exposure to trichloroethylene. Regul Toxicol Pharmacol. 1990 Feb;11(1):24-41. doi: 10.1016/0273-2300(90)90005-v. PMID 2184464
- [Background] Steinberg AD, DeSesso JM. Have animal data been used inappropriately to estimate risks to humans from environmental trichloroethylene? Regul Toxicol Pharmacol. 1993 Oct;18(2):137-53. doi: 10.1006/rtph.1993.1049. PMID 8278637
- [Background] Nelson MA, Bull RJ. Induction of strand breaks in DNA by trichloroethylene and metabolites in rat and mouse liver in vivo. Toxicol Appl Pharmacol. 1988 Jun 15;94(1):45-54. doi: 10.1016/0041-008x(88)90335-3. PMID 3376113
- [Background] Larson JL, Bull RJ. Species differences in the metabolism of trichloroethylene to the carcinogenic metabolites trichloroacetate and dichloroacetate. Toxicol Appl Pharmacol. 1992 Aug;115(2):278-85. doi: 10.1016/0041-008x(92)90333-n. PMID 1641861
- [Background] Henschler D. Metabolism and mutagenicity of halogenated olefins--a comparison of structure and activity. Environ Health Perspect. 1977 Dec;21:61-4. doi: 10.1289/ehp.772161. PMID 348459
- [Background] Buben JA, O'Flaherty EJ. Delineation of the role of metabolism in the hepatotoxicity of trichloroethylene and perchloroethylene: a dose-effect study. Toxicol Appl Pharmacol. 1985 Mar 30;78(1):105-22. doi: 10.1016/0041-008x(85)90310-2. PMID 2994252
- [Background] Bruckner JV, Davis BD, Blancato JN. Metabolism, toxicity, and carcinogenicity of trichloroethylene. Crit Rev Toxicol. 1989;20(1):31-50. doi: 10.3109/10408448909037475. PMID 2673291
- [Background] Van Duuren BL, Banerjee S. Covalent interaction of metabolites of the carcinogen trichloroethylene in rat hepatic microsomes. Cancer Res. 1976 Jul;36(7 PT 1):2419-22. PMID 1277148
- [Background] Henschler D, Romen W, Elsasser HM, Reichert D, Eder E, Radwan Z. Carcinogenicity study of trichloroethylene by longterm inhalation in three animal species. Arch Toxicol. 1980 Feb;43(4):237-48. doi: 10.1007/BF00366179. PMID 7387385
- [Background] Elcombe CR. Species differences in carcinogenicity and peroxisome proliferation due to trichloroethylene: a biochemical human hazard assessment. Arch Toxicol Suppl. 1985;8:6-17. doi: 10.1007/978-3-642-69928-3_2. PMID 3868383
- [Background] Forkert PG, Lash LH, Nadeau V, Tardif R, Simmonds A. Metabolism and toxicity of trichloroethylene in epididymis and testis. Toxicol Appl Pharmacol. 2002 Aug 1;182(3):244-54. doi: 10.1006/taap.2002.9421. PMID 12183104
- [Background] Xu H, Tanphaichitr N, Forkert PG, Anupriwan A, Weerachatyanukul W, Vincent R, Leader A, Wade MG. Exposure to trichloroethylene and its metabolites causes impairment of sperm fertilizing ability in mice. Toxicol Sci. 2004 Dec;82(2):590-7. doi: 10.1093/toxsci/kfh277. Epub 2004 Sep 16. PMID 15375293
- [Background] Gilbert KM, Whitlow AB, Pumford NR. Environmental contaminant and disinfection by-product trichloroacetaldehyde stimulates T cells in vitro. Int Immunopharmacol. 2004 Jan;4(1):25-36. doi: 10.1016/j.intimp.2003.10.001. PMID 14975357
- [Background] Reif JS, Burch JB, Nuckols JR, Metzger L, Ellington D, Anger WK. Neurobehavioral effects of exposure to trichloroethylene through a municipal water supply. Environ Res. 2003 Nov;93(3):248-58. doi: 10.1016/s0013-9351(03)00131-2. PMID 14615234
- [Background] Guehl D, Bezard E, Dovero S, Boraud T, Bioulac B, Gross C. Trichloroethylene and parkinsonism: a human and experimental observation. Eur J Neurol. 1999 Sep;6(5):609-11. doi: 10.1046/j.1468-1331.1999.650609.x. PMID 10457397
- [Background] Miller JW, Uden PC. Characterization of nonvolatile aqueous chlorination products of humic substances. Environ Sci Technol. 1983 Mar 1;17(3):150-7. doi: 10.1021/es00109a006. No abstract available. PMID 22263679
- [Background] Uden PCC, Miller JW. Chlorinated acids and chloral in drinking water. J Amer Water Works Assoc 75:524-527, 1983.
- [Background] Mughal FH. Chlorination of drinking water and cancer: a review. J Environ Pathol Toxicol Oncol. 1992 Sep-Oct;11(5-6):287-92. No abstract available. PMID 1464809
- [Background] Jolley RL. Basic issues in water chlorination: a chemical perspective. In, Water chlorination: chemistry, environmental impact and health effects. Lewis Publ, Inc. Chelsea, MI 5:19-38, 1985.
- [Background] Stacpoole PW. The pharmacology of dichloroacetate. Metabolism. 1989 Nov;38(11):1124-44. doi: 10.1016/0026-0495(89)90051-6. PMID 2554095
- [Background] Abbas RR, Seckel CS, Kidney JK, Fisher JW. Pharmacokinetic analysis of chloral hydrate and its metabolism in B6C3F1 mice. Drug Metab Dispos. 1996 Dec;24(12):1340-6. PMID 8971140
- [Background] Duncan GE, Perkins LA, Theriaque DW, Neiberger RE, Stacpoole PW. Dichloroacetate therapy attenuates the blood lactate response to submaximal exercise in patients with defects in mitochondrial energy metabolism. J Clin Endocrinol Metab. 2004 Apr;89(4):1733-8. doi: 10.1210/jc.2003-031684. PMID 15070938
- [Background] Stacpoole PW, Kerr DS, Barnes C, Bunch ST, Carney PR, Fennell EM, Felitsyn NM, Gilmore RL, Greer M, Henderson GN, Hutson AD, Neiberger RE, O'Brien RG, Perkins LA, Quisling RG, Shroads AL, Shuster JJ, Silverstein JH, Theriaque DW, Valenstein E. Controlled clinical trial of dichloroacetate for treatment of congenital lactic acidosis in children. Pediatrics. 2006 May;117(5):1519-31. doi: 10.1542/peds.2005-1226. PMID 16651305
- [Background] Kaufmann P, Engelstad K, Wei Y, Jhung S, Sano MC, Shungu DC, Millar WS, Hong X, Gooch CL, Mao X, Pascual JM, Hirano M, Stacpoole PW, DiMauro S, De Vivo DC. Dichloroacetate causes toxic neuropathy in MELAS: a randomized, controlled clinical trial. Neurology. 2006 Feb 14;66(3):324-30. doi: 10.1212/01.wnl.0000196641.05913.27. PMID 16476929
- [Background] Salmon AG, Jackson RJ, Smith MT. Chloral hydrate: cancer risk assessment of a drug previously presumed safe. The Toxicologist 11:350, 1991.
- [Background] Liebreich O. Das Chloral hydrat, ein neues Hypnoticum und Anaestheticum, 3rd ed. Berlin: Otto Mullers Verlag, 1869.
- [Background] Reimche LD, Sankaran K, Hindmarsh KW, Kasian GF, Gorecki DK, Tan L. Chloral hydrate sedation in neonates and infants--clinical and pharmacologic considerations. Dev Pharmacol Ther. 1989;12(2):57-64. PMID 2714158
- [Background] Hartley S, Franck LS, Lundergan F. Maintenance sedation of agitated infants in the neonatal intensive care unit with chloral hydrate: new concerns. J Perinatol. 1989 Jun;9(2):162-4. No abstract available. PMID 2738727
- [Background] Krsek P, Sebronova V, Prochazka T, Maulisova A, Komarek V. Successful treatment of Ohtahara syndrome with chloral hydrate. Pediatr Neurol. 2002 Nov;27(5):388-91. doi: 10.1016/s0887-8994(02)00464-2. PMID 12504208
- [Background] Greenberg SB, Faerber EN, Aspinall CL. High dose chloral hydrate sedation for children undergoing CT. J Comput Assist Tomogr. 1991 May-Jun;15(3):467-9. doi: 10.1097/00004728-199105000-00023. PMID 2026812
- [Background] Nathan JE. Management of the refractory young child with chloral hydrate: dosage selection. ASDC J Dent Child. 1987 Mar-Apr;54(2):93-100. PMID 3470333
- [Background] Kuhn JP. CT of the body in children. Pediatr Ann. 1986 May;15(5):367, 371-3, 376-82. doi: 10.3928/0090-4481-19860501-07. PMID 3714334
- [Background] Weir MR, Segapeli JH, Tremper LJ. Sedation for pediatric procedures. Mil Med. 1986 Mar;151(3):181-4. No abstract available. PMID 3085006
- [Background] Miller RR, Greenblatt DJ. Clinical effects of chloral hydrate in hospitalized medical patients. J Clin Pharmacol. 1979 Oct;19(10):669-74. doi: 10.1002/j.1552-4604.1979.tb01630.x. No abstract available. PMID 512063
- [Background] Malviya S, Voepel-Lewis T, Tait AR, Reynolds PI, Gujar SK, Gebarski SS, Petter Eldevik O. Pentobarbital vs chloral hydrate for sedation of children undergoing MRI: efficacy and recovery characteristics. Paediatr Anaesth. 2004 Jul;14(7):589-95. doi: 10.1111/j.1460-9592.2004.01243.x. PMID 15200658
- [Background] James MO, Cornett R, Yan Z, Henderson GN, Stacpoole PW. Glutathione-dependent conversion to glyoxylate, a major pathway of dichloroacetate biotransformation in hepatic cytosol from humans and rats, is reduced in dichloroacetate-treated rats. Drug Metab Dispos. 1997 Nov;25(11):1223-7. PMID 9351896
- [Background] Cornett R, James MO, Henderson GN, Cheung J, Shroads AL, Stacpoole PW. Inhibition of glutathione S-transferase zeta and tyrosine metabolism by dichloroacetate: a potential unifying mechanism for its altered biotransformation and toxicity. Biochem Biophys Res Commun. 1999 Sep 7;262(3):752-6. doi: 10.1006/bbrc.1999.1287. PMID 10471397
- [Background] Tong Z, Board PG, Anders MW. Glutathione transferase zeta catalyses the oxygenation of the carcinogen dichloroacetic acid to glyoxylic acid. Biochem J. 1998 Apr 15;331 ( Pt 2)(Pt 2):371-4. doi: 10.1042/bj3310371. PMID 9531472
- [Background] Fernandez-Canon JM, Hejna J, Reifsteck C, Olson S, Grompe M. Gene structure, chromosomal location, and expression pattern of maleylacetoacetate isomerase. Genomics. 1999 Jun 15;58(3):263-9. doi: 10.1006/geno.1999.5832. PMID 10373324
- [Background] Blackburn AC, Coggan M, Tzeng HF, Lantum H, Polekhina G, Parker MW, Anders MW, Board PG. GSTZ1d: a new allele of glutathione transferase zeta and maleylacetoacetate isomerase. Pharmacogenetics. 2001 Nov;11(8):671-8. doi: 10.1097/00008571-200111000-00005. PMID 11692075
- [Background] Blackburn AC, Tzeng HF, Anders MW, Board PG. Discovery of a functional polymorphism in human glutathione transferase zeta by expressed sequence tag database analysis. Pharmacogenetics. 2000 Feb;10(1):49-57. doi: 10.1097/00008571-200002000-00007. PMID 10739172
- [Background] MARSHALL EK Jr, OWENS AH Jr. Absorption, excretion and metabolic fate of chloral hydrate and trichloroethanol. Bull Johns Hopkins Hosp. 1954 Jul;95(1):1-18. No abstract available. PMID 13172552
- [Background] Jochemsen R, Breimer DD. Pharmacokinetics of benzodiazepines: metabolic pathways and plasma level profiles. Curr Med Res Opin. 1984;8 Suppl 4:60-79. doi: 10.1185/03007998409109545. PMID 6144464
- [Background] Henderson GN, Yan Z, James MO, Davydova N, Stacpoole PW. Kinetics and metabolism of chloral hydrate in children: identification of dichloroacetate as a metabolite. Biochem Biophys Res Commun. 1997 Jun 27;235(3):695-8. doi: 10.1006/bbrc.1997.6868. PMID 9207222
- [Background] Toxicological review of dichloroacetic acid (CAS No. 79-43-6). U.S. Environ. Protection Agency. Washington, DC, August, 2003.
- [Background] Bull RJ, Sanchez IM, Nelson MA, Larson JL, Lansing AJ. Liver tumor induction in B6C3F1 mice by dichloroacetate and trichloroacetate. Toxicology. 1990 Sep;63(3):341-59. doi: 10.1016/0300-483x(90)90195-m. PMID 2219130
- [Background] Daniel FB, DeAngelo AB, Stober JA, Olson GR, Page NP. Hepatocarcinogenicity of chloral hydrate, 2-chloroacetaldehyde, and dichloroacetic acid in the male B6C3F1 mouse. Fundam Appl Toxicol. 1992 Aug;19(2):159-68. doi: 10.1016/0272-0590(92)90147-a. PMID 1516771
- [Background] DeAngelo AB, Daniel FB, Stober JA, Olson GR. The carcinogenicity of dichloroacetic acid in the male B6C3F1 mouse. Fundam Appl Toxicol. 1991 Feb;16(2):337-47. doi: 10.1016/0272-0590(91)90118-n. PMID 2055364
- [Background] Pereira MA, Li K, Kramer PM. Promotion by mixtures of dichloroacetic acid and trichloroacetic acid of N-methyl-N-nitrosourea-initiated cancer in the liver of female B6C3F1 mice. Cancer Lett. 1997 May 1;115(1):15-23. doi: 10.1016/s0304-3835(97)04699-5. PMID 9097974
- [Background] Pereira MA, Phelps JB. Promotion by dichloroacetic acid and trichloroacetic acid of N-methyl-N-nitrosourea-initiated cancer in the liver of female B6C3F1 mice. Cancer Lett. 1996 Apr 19;102(1-2):133-41. doi: 10.1016/0304-3835(96)04156-0. PMID 8603361
- [Background] DeAngelo AB, Daniel FB, Most BM, Olson GR. The carcinogenicity of dichloroacetic acid in the male Fischer 344 rat. Toxicology. 1996 Dec 18;114(3):207-21. doi: 10.1016/s0300-483x(96)03510-x. PMID 8980710
- [Background] McHugh Law J, Lopez L, DeAngelo AB. Hepatotoxicity of the drinking water disinfection by-product, dichloroacetic acid, in the medaka small fish model. Toxicol Lett. 1998 Jan 16;94(1):19-27. doi: 10.1016/s0378-4274(97)00095-7. PMID 9544695
- [Background] Kato-Weinstein J, Lingohr MK, Orner GA, Thrall BD, Bull RJ. Effects of dichloroacetate on glycogen metabolism in B6C3F1 mice. Toxicology. 1998 Sep 15;130(2-3):141-54. doi: 10.1016/s0300-483x(98)00106-1. PMID 9865481
- [Background] Stacpoole PW, Henderson GN, Yan Z, Cornett R, James MO. Pharmacokinetics, metabolism and toxicology of dichloroacetate. Drug Metab Rev. 1998 Aug;30(3):499-539. doi: 10.3109/03602539808996323. No abstract available. PMID 9710704
- [Background] DeAngelo AB, Daniel FB, McMillan L, Wernsing P, Savage RE Jr. Species and strain sensitivity to the induction of peroxisome proliferation by chloroacetic acids. Toxicol Appl Pharmacol. 1989 Nov;101(2):285-98. doi: 10.1016/0041-008x(89)90277-9. PMID 2815084
- [Background] Everhart JL, Kurtz DT, McMillan JM. Dichloroacetic acid induction of peroxisome proliferation in cultured hepatocytes. J Biochem Mol Toxicol. 1998;12(6):351-9. doi: 10.1002/(sici)1099-0461(1998)12:63.0.co;2-2. PMID 9736484
- [Background] Zhou YC, Waxman DJ. Activation of peroxisome proliferator-activated receptors by chlorinated hydrocarbons and endogenous steroids. Environ Health Perspect. 1998 Aug;106 Suppl 4(Suppl 4):983-8. doi: 10.1289/ehp.98106s4983. PMID 9703482
- [Background] Maloney EK, Waxman DJ. trans-Activation of PPARalpha and PPARgamma by structurally diverse environmental chemicals. Toxicol Appl Pharmacol. 1999 Dec 1;161(2):209-18. doi: 10.1006/taap.1999.8809. PMID 10581215
- [Background] Sanchez IM, Bull RJ. Early induction of reparative hyperplasia in the liver of B6C3F1 mice treated with dichloroacetate and trichloroacetate. Toxicology. 1990 Oct;64(1):33-46. doi: 10.1016/0300-483x(90)90097-z. PMID 2219131
- [Background] Snyder RD, Pullman J, Carter JH, Carter HW, DeAngelo AB. In vivo administration of dichloroacetic acid suppresses spontaneous apoptosis in murine hepatocytes. Cancer Res. 1995 Sep 1;55(17):3702-5. PMID 7641179
- [Background] Lingohr MK, Thrall BD, Bull RJ. Effects of dichloroacetate (DCA) on serum insulin levels and insulin-controlled signaling proteins in livers of male B6C3F1 mice. Toxicol Sci. 2001 Jan;59(1):178-84. doi: 10.1093/toxsci/59.1.178. PMID 11134557
- [Background] Gonzalez-Leon A, Schultz IR, Bull RJ. Species differences in the toxicokinetics of dichloroacetate and trichloroacetate in F344 rats and B6C3F1 mice after prolonged administration in drinking water. Fundam Appl Toxicol Suppl 36, Abst. 168, p. 33, 1997.
- [Background] Gonzalez-Leon A, Schultz IR, Xu G, Bull RJ. Pharmacokinetics and metabolism of dichloroacetate in the F344 rat after prior administration in drinking water. Toxicol Appl Pharmacol. 1997 Oct;146(2):189-95. doi: 10.1006/taap.1997.8232. PMID 9344886
- [Background] Waxman DJ. P450 gene induction by structurally diverse xenochemicals: central role of nuclear receptors CAR, PXR, and PPAR. Arch Biochem Biophys. 1999 Sep 1;369(1):11-23. doi: 10.1006/abbi.1999.1351. PMID 10462436
- [Background] DeMarini DM, Perry E, Shelton ML. Dichloroacetic acid and related compounds: induction of prophage in E. coli and mutagenicity and mutation spectra in Salmonella TA100. Mutagenesis. 1994 Sep;9(5):429-37. doi: 10.1093/mutage/9.5.429. PMID 7837977
- [Background] Fox AW, Yang X, Murli H, Lawlor TE, Cifone MA, Reno FE. Absence of mutagenic effects of sodium dichloroacetate. Fundam Appl Toxicol. 1996 Jul;32(1):87-95. doi: 10.1006/faat.1996.0110. PMID 8812237
- [Background] Fuscoe JC, Afshari AJ, George MH, DeAngelo AB, Tice RR, Salman T, Allen JW. In vivo genotoxicity of dichloroacetic acid: evaluation with the mouse peripheral blood micronucleus assay and the single cell gel assay. Environ Mol Mutagen. 1996;27(1):1-9. doi: 10.1002/(SICI)1098-2280(1996)27:13.0.CO;2-L. PMID 8625942
- [Background] Giller S, Le Curieux F, Erb F, Marzin D. Comparative genotoxicity of halogenated acetic acids found in drinking water. Mutagenesis. 1997 Sep;12(5):321-8. doi: 10.1093/mutage/12.5.321. PMID 9379909
- [Background] Harrington-Brock K, Doerr CL, Moore MM. Mutagenicity of three disinfection by-products: di- and trichloroacetic acid and chloral hydrate in L5178Y/TK +/- (-)3.7.2C mouse lymphoma cells. Mutat Res. 1998 Mar 30;413(3):265-76. doi: 10.1016/s1383-5718(98)00026-6. PMID 9651541
- [Background] Leavitt SA, DeAngelo AB, George MH, Ross JA. Assessment of the mutagenicity of dichloroacetic acid in lacI transgenic B6C3F1 mouse liver. Carcinogenesis. 1997 Nov;18(11):2101-6. doi: 10.1093/carcin/18.11.2101. PMID 9395208
- [Background] Rapson WH, Nazar MA, Butsky VV. Mutagenicity produced by aqueous chlorination of organic compounds. Bull Environ Contam Toxicol. 1980 Apr;24(4):590-6. doi: 10.1007/BF01608160. No abstract available. PMID 6991030
- [Background] Waskell L. A study of the mutagenicity of anesthetics and their metabolites. Mutat Res. 1978 May;57(2):141-53. doi: 10.1016/0027-5107(78)90261-0. PMID 351387
- [Background] Mariash CN, Schwartz HL. Effect of dichloroacetic acid on rat hepatic messenger RNA activity profiles. Metabolism. 1986 May;35(5):452-6. doi: 10.1016/0026-0495(86)90137-x. PMID 3702676
- [Background] Barton CH, Bailey E. Changes in immunoreactive malic enzyme in liver and brown adipose tissue during development of the rat. J Dev Physiol. 1987 Jun;9(3):215-24. PMID 3611638
- [Background] Barak C, Reed MK, Maniscalco SP, Sherry AD, Malloy CR, Jessen ME. Effects of dichloroacetate on mechanical recovery and oxidation of physiologic substrates after ischemia and reperfusion in the isolated heart. J Cardiovasc Pharmacol. 1998 Mar;31(3):336-44. doi: 10.1097/00005344-199803000-00002. PMID 9514176
- [Background] Stacpoole PW, Harwood HJ Jr, Cameron DF, Curry SH, Samuelson DA, Cornwell PE, Sauberlich HE. Chronic toxicity of dichloroacetate: possible relation to thiamine deficiency in rats. Fundam Appl Toxicol. 1990 Feb;14(2):327-37. doi: 10.1016/0272-0590(90)90212-3. PMID 2318357
- [Background] Hong JY, Pan JM, Gonzalez FJ, Gelboin HV, Yang CS. The induction of a specific form of cytochrome P-450 (P-450j) by fasting. Biochem Biophys Res Commun. 1987 Feb 13;142(3):1077-83. doi: 10.1016/0006-291x(87)91525-7. PMID 3827895
- [Background] Yoo JS, Park HS, Ning SM, Lee MJ, Yang CS. Effects of thiamine deficiency on hepatic cytochromes P450 and drug-metabolizing enzyme activities. Biochem Pharmacol. 1990 Feb 1;39(3):519-25. doi: 10.1016/0006-2952(90)90059-t. PMID 2306264
- [Background] Yang HM, Houser WH, Davis ME. Dichloroacetic acid treatment increases hepatic CYP2E1 in male and female rats. Toxicol Appl Pharmacol. 1996 Dec;141(2):382-8. doi: 10.1006/taap.1996.0303. PMID 8975762
- [Background] Thai SF, Allen JW, DeAngelo AB, George MH, Fuscoe JC. Detection of early gene expression changes by differential display in the livers of mice exposed to dichloroacetic acid. Carcinogenesis. 2001 Aug;22(8):1317-22. doi: 10.1093/carcin/22.8.1317. PMID 11470764
- [Background] NTP Technical Report. Toxicology and carcinogenesis study of chloral hydrate. NIH Publication No. 03-4437, 2002.
- [Background] IARC Monographs on the Evaluation of Carcinogenic Risks to Humans. Chloral hydrate. World Health Organization, 2004, pp. 317-358.
- [Background] Davidson IW, Beliles RP. Consideration of the target organ toxicity of trichloroethylene in terms of metabolite toxicity and pharmacokinetics. Drug Metab Rev. 1991;23(5-6):493-599. doi: 10.3109/03602539109029772. PMID 1802654
- [Background] Ikbal M, Tastekin A, Dogan H, Pirim I, Ors R. The assessment of genotoxic effects in lymphocyte cultures of infants treated with chloral hydrate. Mutat Res. 2004 Dec 12;564(2):159-64. doi: 10.1016/j.mrgentox.2004.08.007. PMID 15507380
- [Background] Ho YS, Ma HY, Chang HY, Wei BL, Lee CC, Ho SY, Guo HR, Wu TP, Chang WH, Wang YJ. Lipid peroxidation and cell death mechanisms in rats and human cells induced by chloral hydrate. Food Chem Toxicol. 2003 May;41(5):621-9. doi: 10.1016/s0278-6915(02)00323-x. PMID 12659714
- [Background] Harinath S, Sikdar SK. Trichloroethanol enhances the activity of recombinant human TREK-1 and TRAAK channels. Neuropharmacology. 2004 Apr;46(5):750-60. doi: 10.1016/j.neuropharm.2003.11.023. PMID 14996553
- [Background] Fischer W, Wirkner K, Weber M, Eberts C, Koles L, Reinhardt R, Franke H, Allgaier C, Gillen C, Illes P. Characterization of P2X3, P2Y1 and P2Y4 receptors in cultured HEK293-hP2X3 cells and their inhibition by ethanol and trichloroethanol. J Neurochem. 2003 May;85(3):779-90. doi: 10.1046/j.1471-4159.2003.01716.x. PMID 12694404
- [Background] Sabeti J, Gerhardt GA, Zahniser NR. Chloral hydrate and ethanol, but not urethane, alter the clearance of exogenous dopamine recorded by chronoamperometry in striatum of unrestrained rats. Neurosci Lett. 2003 May 29;343(1):9-12. doi: 10.1016/s0304-3940(03)00301-x. PMID 12749985
- [Background] Akundi RS, Macho A, Munoz E, Lieb K, Bringmann G, Clement HW, Hull M, Fiebich BL. 1-trichloromethyl-1,2,3,4-tetrahydro-beta-carboline-induced apoptosis in the human neuroblastoma cell line SK-N-SH. J Neurochem. 2004 Oct;91(2):263-73. doi: 10.1111/j.1471-4159.2004.02710.x. PMID 15447660
- [Background] Templin MV, Parker JC, Bull RJ. Relative formation of dichloroacetate and trichloroacetate from trichloroethylene in male B6C3F1 mice. Toxicol Appl Pharmacol. 1993 Nov;123(1):1-8. doi: 10.1006/taap.1993.1214. PMID 8236248
- [Background] Gribble GW. Naturally occurring organohalogen compounds--a comprehensive survey. Fortschr Chem Org Naturst. 1996;68:1-423. No abstract available. PMID 8795309
- [Background] Agbenyega T, Planche T, Bedu-Addo G, Ansong D, Owusu-Ofori A, Bhattaram VA, Nagaraja NV, Shroads AL, Henderson GN, Hutson AD, Derendorf H, Krishna S, Stacpoole PW. Population kinetics, efficacy, and safety of dichloroacetate for lactic acidosis due to severe malaria in children. J Clin Pharmacol. 2003 Apr;43(4):386-96. doi: 10.1177/0091270003251392. PMID 12723459
- [Background] Yan Z, Henderson GN, James MO, Stacpoole PW. Determination of dichloroacetate and its metabolites in human plasma by gas chromatography-mass spectrometry. J Chromatogr B Biomed Sci Appl. 1997 Dec 5;703(1-2):75-84. doi: 10.1016/s0378-4347(97)00404-0. PMID 9448064
- [Background] Jia M, Wu WW, Yost RA, Chadik PA, Stacpoole PW, Henderson GN. Simultaneous determination of trace levels of nine haloacetic acids in biological samples as their pentafluorobenzyl derivatives by gas chromatography/tandem mass spectrometry in electron capture negative ion chemical ionization mode. Anal Chem. 2003 Aug 15;75(16):4065-80. doi: 10.1021/ac034036w. PMID 14632119
- [Background] Stacpoole PW, Moore GW, Kornhauser DM. Toxicity of chronic dichloroacetate. N Engl J Med. 1979 Feb 15;300(7):372. doi: 10.1056/NEJM197902153000726. No abstract available. PMID 215910
- [Background] Stacpoole PW, Barnes CL, Hurbanis MD, Cannon SL, Kerr DS. Treatment of congenital lactic acidosis with dichloroacetate. Arch Dis Child. 1997 Dec;77(6):535-41. doi: 10.1136/adc.77.6.535. No abstract available. PMID 9496194
- [Background] Stacpoole PW, Harman EM, Curry SH, Baumgartner TG, Misbin RI. Treatment of lactic acidosis with dichloroacetate. N Engl J Med. 1983 Aug 18;309(7):390-6. doi: 10.1056/NEJM198308183090702. PMID 6877297
- [Background] Stacpoole PW, Moore GW, Kornhauser DM. Metabolic effects of dichloroacetate in patients with diabetes mellitus and hyperlipoproteinemia. N Engl J Med. 1978 Mar 9;298(10):526-30. doi: 10.1056/NEJM197803092981002. PMID 625308
- [Background] Neiberger RE, George JC, Perkins LA, Theriaque DW, Hutson AD, Stacpoole PW. Renal manifestations of congenital lactic acidosis. Am J Kidney Dis. 2002 Jan;39(1):12-23. doi: 10.1053/ajkd.2002.29872. PMID 11774096
- [Background] Ammini CV, Fernandez-Canon J, Shroads AL, Cornett R, Cheung J, James MO, Henderson GN, Grompe M, Stacpoole PW. Pharmacologic or genetic ablation of maleylacetoacetate isomerase increases levels of toxic tyrosine catabolites in rodents. Biochem Pharmacol. 2003 Nov 15;66(10):2029-38. doi: 10.1016/j.bcp.2003.07.002. PMID 14599561
- [Background] Guo X, Dixit V, Liu H, Shroads AL, Henderson GN, James MO, Stacpoole PW. Inhibition and recovery of rat hepatic glutathione S-transferase zeta and alteration of tyrosine metabolism following dichloroacetate exposure and withdrawal. Drug Metab Dispos. 2006 Jan;34(1):36-42. doi: 10.1124/dmd.105.003996. Epub 2005 Sep 30. PMID 16199472
- [Background] Holme E, Lindstedt S. Tyrosinaemia type I and NTBC (2-(2-nitro-4-trifluoromethylbenzoyl)-1,3-cyclohexanedione). J Inherit Metab Dis. 1998 Aug;21(5):507-17. doi: 10.1023/a:1005410820201. PMID 9728331
- [Background] Fujita H, Koizumi A, Yamamoto M, Kumai M, Sadamoto T, Ikeda M. Inhibition of delta-aminolevulinate dehydratase in trichloroethylene-exposed rats, and the effects on heme regulation. Biochim Biophys Acta. 1984 Jul 16;800(1):1-10. doi: 10.1016/0304-4165(84)90087-4. PMID 6743680
- [Background] Grompe M, Overturf K, al-Dhalimy M, Finegold M. Therapeutic trials in the murine model of hereditary tyrosinaemia type I: a progress report. J Inherit Metab Dis. 1998 Aug;21(5):518-31. doi: 10.1023/a:1005462804271. PMID 9728332
- [Background] Grompe M, Lindstedt S, al-Dhalimy M, Kennaway NG, Papaconstantinou J, Torres-Ramos CA, Ou CN, Finegold M. Pharmacological correction of neonatal lethal hepatic dysfunction in a murine model of hereditary tyrosinaemia type I. Nat Genet. 1995 Aug;10(4):453-60. doi: 10.1038/ng0895-453. PMID 7545495
- [Background] Fernandez-Canon JM, Baetscher MW, Finegold M, Burlingame T, Gibson KM, Grompe M. Maleylacetoacetate isomerase (MAAI/GSTZ)-deficient mice reveal a glutathione-dependent nonenzymatic bypass in tyrosine catabolism. Mol Cell Biol. 2002 Jul;22(13):4943-51. doi: 10.1128/MCB.22.13.4943-4951.2002. PMID 12052898
- [Background] Shroads AL, Henderson GN, Cheung J, James MO, Stacpoole PW. Unified gas chromatographic-mass spectrometric method for quantitating tyrosine metabolites in urine and plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Sep 5;808(2):153-61. doi: 10.1016/j.jchromb.2004.05.005. PMID 15261808
- [Background] Felitsyn NM, Henderson GN, James MO, Stacpoole PW. Liquid chromatography-tandem mass spectrometry method for the simultaneous determination of delta-ALA, tyrosine and creatinine in biological fluids. Clin Chim Acta. 2004 Dec;350(1-2):219-30. doi: 10.1016/j.cccn.2004.08.009. PMID 15530481
- [Background] Tzeng HF, Blackburn AC, Board PG, Anders MW. Polymorphism- and species-dependent inactivation of glutathione transferase zeta by dichloroacetate. Chem Res Toxicol. 2000 Apr;13(4):231-6. doi: 10.1021/tx990175q. PMID 10775321
- [Background] Anderson WB, Liebler DC, Board PG, Anders MW. Mass spectral characterization of dichloroacetic acid-modified human glutathione transferase zeta. Chem Res Toxicol. 2002 Nov;15(11):1387-97. doi: 10.1021/tx025553x. PMID 12437329
- [Background] Anderson WB, Board PG, Anders MW. Glutathione transferase zeta-catalyzed bioactivation of dichloroacetic acid: reaction of glyoxylate with amino acid nucleophiles. Chem Res Toxicol. 2004 May;17(5):650-62. doi: 10.1021/tx034099+. PMID 15144222
- [Background] Kinter M, Sherman NE. Peptide Sequencng andIdentifcation Using Tandem Mass Specrometry. John Wiley and Sons, Inc., pp. 147-165, 2000.
- [Background] Cohen SL, Chait BT. Mass spectrometry of whole proteins eluted from sodium dodecyl sulfate-polyacrylamide gel electrophoresis gels. Anal Biochem. 1997 May 1;247(2):257-67. doi: 10.1006/abio.1997.2072. PMID 9177686
- [Background] LoPachin RM, Jones RC, Patterson TA, Slikker W Jr, Barber DS. Application of proteomics to the study of molecular mechanisms in neurotoxicology. Neurotoxicology. 2003 Dec;24(6):761-75. doi: 10.1016/j.neuro.2003.08.003. PMID 14637371
- [Background] Righetti PG, Castagna A, Antonucci F, Piubelli C, Cecconi D, Campostrini N, Zanusso G, Monaco S. The proteome: anno Domini 2002. Clin Chem Lab Med. 2003 Apr;41(4):425-38. doi: 10.1515/CCLM.2003.065. PMID 12747583
- [Background] Gygi SP, Rist B, Gerber SA, Turecek F, Gelb MH, Aebersold R. Quantitative analysis of complex protein mixtures using isotope-coded affinity tags. Nat Biotechnol. 1999 Oct;17(10):994-9. doi: 10.1038/13690. PMID 10504701
- [Background] Proteome Research: mass spectrometry. Peter James. Springer, pp. 5-9 2001.
- [Background] Nguyen MH, Keeffe EB. Chronic hepatitis B and hepatitis C in Asian Americans. Rev Gastroenterol Disord. 2003 Summer;3(3):125-34. PMID 14502116
- [Background] Mortazavi B, Chanton JP. A rapid and precise technique for measuring delta(13)C-CO(2) and delta(18)O-CO(2) ratios at ambient CO(2) concentrations for biological applications and the influence of container type and storage time on the sample isotope ratios. Rapid Commun Mass Spectrom. 2002;16(14):1398-403. doi: 10.1002/rcm.730. PMID 12112620
- [Background] Ronaghi M. Pyrosequencing sheds light on DNA sequencing. Genome Res. 2001 Jan;11(1):3-11. doi: 10.1101/gr.11.1.3. PMID 11156611
- [Background] Ritz MA, Fraser R, Edwards N, Di Matteo AC, Chapman M, Butler R, Cmielewski P, Tournadre JP, Davidson G, Dent J. Delayed gastric emptying in ventilated critically ill patients: measurement by 13 C-octanoic acid breath test. Crit Care Med. 2001 Sep;29(9):1744-9. doi: 10.1097/00003246-200109000-00015. PMID 11546976
- [Background] Stacpoole PW, Wright EC, Baumgartner TG, Bersin RM, Buchalter S, Curry SH, Duncan CA, Harman EM, Henderson GN, Jenkinson S, et al. A controlled clinical trial of dichloroacetate for treatment of lactic acidosis in adults. The Dichloroacetate-Lactic Acidosis Study Group. N Engl J Med. 1992 Nov 26;327(22):1564-9. doi: 10.1056/NEJM199211263272204. PMID 1435883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited by a posted advertisement.
Pre-assignment Details: Two subjects were enrolled but did not participate in the study. One subject was delayed because the solution for the infusion had particles in it and then didn't continue(didn't receive any intervention) due to funding issues, and the second one was enrolled but didn't receive any intervention due to funding issues that have been explained.
Period: Overall Study
Arm/Group | Haplotypes and DCA Metabolism
Started | 2
Completed | 0
Not Completed | 2
Not completed — Infusion cost exceeded funding | 2

BASELINE CHARACTERISTICS:
Arm/Group | Haplotypes and DCA Metabolism
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: The Interaction of DCA and/or Tyrosine Breakdown Products and Maleylacetoacetate Isomerase (MAAI) in Vivo.
Description: Subjects are administered an infusion of the amino acids leucine and tyrosine. The next day they start a five day course of dichloroacetate(DCA). At the end of five days they receive another infusion of tyrosine and leucine.
  The pharmacokinetics of DCA is calculated following the second infusion.
Time Frame: One week
Population: No statistical analysis. The data was incomplete and was not analyzed.
Groups:
- The Interaction of DCA and/or Tyrosine Breakdown Products: Healthy men and women with different haplotypes will receive an infusion of leucine and tyrosine. The following day they begin a 5 day course of dichloroacetate (DCA)at a dose of 2.5mcg/kg/day. On day 6 they return and receive another infusion of leucine and tyrosine. After a 30 day washout period the subject returns and again receives an infusion of leucine and tyrosine. Then on day 2 they begin a dose of DCA at 25mg/kg for 5 days and then return for the final infusion of leucine and tyrosine.
Arm/Group | The Interaction of DCA and/or Tyrosine Breakdown Products
Number analyzed (Participants) | 0

2. Secondary Outcome: Inhibition of Tyrosine and Individual's Haplotype
Description: Given the infusion of the above amino acids and DCA administration the inhibition of tyrosine will be measured in the KRT haplotype and non KRT haplotype.
Time Frame: one week
Population: No statistical analysis. The data was incomplete and was not analyzed.
Arm/Group | Haplotypes and DCA Metabolism
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: August 2011 to January 2012
Arm/Group | Haplotypes and DCA Metabolism
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haplotypes and DCA Metabolism (N=2)
dizziness (Nervous system disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1) — Patient fainted for 15 seconds when blood was drawn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No